CLINICAL TRIAL: NCT05995119
Title: A Phase I, Randomized, Single-Dose, Open-Label, Four-Way Crossover Study to Evaluate the Comparative Bioavailability of Apixaban for TAH3311 Oral Dissolving Film Versus ELIQUIS® Oral Tablet in Healthy Male and Female Subjects
Brief Title: Comparative Bioavailability Study of TAH3311 5 mg Oral Dissolving Film vs ELIQUIS® 5 mg Tablet in Healthy Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: TAHO Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: TAH3311-12288201
Record Dates: First submitted 2023-07-24; First posted 2023-08-16 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Healthy Volunteers; Fasting; Fed
MeSH Terms: conditions — Fasting; Lecithin Cholesterol Acyltransferase Deficiency | interventions — apixaban; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Comparative Bioavailability of apixaban film (TAH3311) and Eliquis Tablet in fed conditions (Other)
  Interventions: Drug: Apixaban 5 mg Oral Dissolving Film (TAH3311) and Tablet (Eliquis®)
- Comparative Bioavailability of apixaban film (TAH3311) and Eliquis Tablet in fast conditions (Other)
  Interventions: Drug: Apixaban 5 mg Oral Dissolving Film (TAH3311) and Tablet (Eliquis®)

INTERVENTIONS:
Drug: Apixaban 5 mg Oral Dissolving Film (TAH3311) and Tablet (Eliquis®) — The subjects were administered either the test (TAH3311 5 mg ODF as Treatment T1) or reference (ELIQUIS® 5 mg oral tablet as Treatment R1) product at 30 minutes following the start of a standardized high-fat, high-calorie breakfast that was preceded by an overnight fast of at least 10 hours. In the other two study periods, the subjects were administered either the test (Treatment T2) or reference (Treatment R2) product following an overnight fast of at least 10 hours. The subjects received the test and reference products in accordance with a four-sequence randomization schedule. There was a washout period of 5 days between the dosing days of any two consecutive periods.
  Other Names: TAH3311 5 mg ODF

SUMMARY:
The goal of this clinical trial is to evaluate the pharmacokinetic profiles and bioequivalence, and to determine the safety and tolerability of the TAH3311 Oral Dissolving Film (ODF) 5mg compared with ELIQUIS® (Apixaban) 5mg Oral Tablet, after single dose under fasted and fed conditions in healthy volunteers.

DETAILED DESCRIPTION:
For Treatment T1, the test product was administered orally at 30 minutes after the start of a standardized high-fat, high-calorie breakfast that was preceded by an overnight fast of at least 10 hours. For Treatment T2, the test product was administered orally following an overnight fast of at least 10 hours.

The test treatment (1 × TAH3311 (apixaban) oral dissolving film 5 mg) was placed on the top of the tongue. Subjects were asked to close their mouth naturally and not to swallow for at least 60 seconds or until they felt that the film had fully dissolved. They were asked to indicate this to the dosing staff by raising their hand, who then verified. If any film remained in the mouth, after the subject raised his/her hand, the subject was reminded to not swallow and requested to close their mouth and allow the film to continue to dissolve and the study staff monitored the subject's mouth every 1 minute until such time that the film had fully dissolved. The time taken from dosing until the film had completely dissolved was documented. Dosing time was considered the time when the film was placed on the subject's tongue.

No water was administered with the Test Treatments (T1 and T2).

Reference Treatments (R1 & R2):

For Treatment R1, the reference product was administered orally at 30 minutes after the start of a standardized high-fat, high-calorie breakfast that was preceded by an overnight fast of at least 10 hours. For Treatment R2, the reference product was administered orally following an overnight fast of at least 10 hours.

Each dose was administered with 240 mL of room temperature water. Subjects were instructed to swallow the tablet whole without chewing or biting. Any subject, who bit or chewed the tablet, was dropped from the study. Immediately after dosing a mouth check was performed to ensure that the tablet was swallowed whole without chewing or biting.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant, non-lactating females, 18-80 years of age, inclusive.
2. A minimum body weight of 60 kg and a Body Mass Index (BMI) of 18.5-29.9 kg/m², inclusive. BMI will be calculated using Novum Pharmaceutical Research Services Standard Operating Procedures.
3. Female subjects must meet at least one of the following requirements:

   * Agree to abstain from sexual intercourse from screening and throughout the duration of the study, including washout periods, and for 30 days after the last study drug administration.
   * Have used and agree to continue to use a reliable method of hormonal contraception (oral, implanted, or injected) in conjunction with a barrier method (e.g., diaphragm, cervical cap, male condom, and female condom and spermicidal foam, sponges, and film) for at least 30 days before initial dosing and throughout the duration of the study, including washout periods, and for 30 days after the last study drug administration.
   * Have used and agree to continue to use an intrauterine device (IUD) at least 3 months before initial dosing and throughout the duration of the study, including washout periods, and for 30 days after the last study drug administration.
   * Surgically sterile (bilateral oophorectomy or hysterectomy, bilateral tubal ligation at least 3 months before initial dosing or Essure® device placement before the year 2018).
   * At least 2 years postmenopausal and have a documented follicle stimulating hormone (FSH) level ≥ 40 milli-international units per milliliter (mIU/mL) at screening.
4. Male subjects who are not surgically sterile must agree to abstain from sexual intercourse (complete abstinence) or use appropriate contraceptive measures and agree to not impregnate a female partner(s) and not to donate sperm throughout the entire study, including the washout periods, and for 30 days after the last study drug administration. Examples of acceptable methods of contraception include a double-barrier method of contraception (e.g., condom with spermicide). Other forms of contraception may be acceptable, at the discretion of the Investigator.
5. Subject is judged by an Investigator to be in good health as determined by lack of clinically significant abnormalities in health assessments performed at screening. Any abnormalities or deviations outside the normal ranges for any clinical testing (e.g., laboratory tests, ECG, vital signs) may be repeated, at the discretion of the Investigator(s), and judged by an Investigator to be not clinically significant for study participation.
6. Subject doesn't have any relevant dietary restrictions, as determined by the Investigator, and is willing to consume a high-fat, high-calorie breakfast and other standard meals provided during the treatment periods of the study, and to comply with the fasting conditions required by the study design.
7. Subject is able to read and speak English fluently. Subjects will be required to read, understand, sign and date the informed consent form, which meets all criteria of current FDA regulations, and must be able to understand the information and instruction given to them during the study.

Exclusion Criteria:

1. Females who are pregnant, lactating, or likely to become pregnant during the study.
2. History of allergy or sensitivity to apixaban, or history of any food or drug hypersensitivity or intolerance which, in the opinion of the Investigator, would compromise the safety of the subject or the study.
3. Current tongue piercing or other piercings in the mouth, including lips and cheeks which have studs/rings, etc. or where the piercing wound is not completely closed or any tongue or other oral deformities that may affect the absorption of the drug product.
4. Significant history or current evidence of system disorders, organ dysfunction especially cardiovascular disorders (e.g., atrial fibrillation), renal or hepatic disorders.
5. Significant familial history of sudden cardiac death, as determined by the Investigator.
6. Subject has a prosthetic heart valve.
7. Significant history or current evidence of blood clots or bleeding disorders (e.g., bleeding diathesis [tendency to bleed or bruise easily]), stroke, or active pathological bleeding.
8. Clinically significant history or are currently at risk for arterial or venous thromboembolic events (e.g., transient ischemic attack, cerebrovascular accident, myocardial infarction, retinal artery occlusion or retinal vein thrombosis, pulmonary embolism, deep vein thrombosis, antiphospholipid syndrome), as determined by the Investigator.
9. Serum creatinine ≥ 1.5 mg/dL.
10. Creatinine clearance (CrCl) < 50 mL/min; obtained from the clinical laboratory tests performed at screening. CrCl can be estimated using the following (Cockcroft-Gault) equation:

    CrCl= ((140-age) × actual weight(kg) × [0.85 if female])/(SerumCr(mg⁄dL) × 72)
11. Clinically significant history or presence of gastrointestinal disease (e.g., bleeding, perforation, or fistulas) or malabsorption, as determined by the Investigator.
12. Subject has had an acute infection within 2 weeks before screening or at any time between screening and check-in including, but not limited to, history, signs, or symptoms of a common cold (e.g., mild rhinorrhea), untreated oral/dental abnormalities (e.g., untreated dental caries as determined by examination of the mouth), or untreated disruption of the skin, as determined by the Investigator.
13. Subject has an active infection requiring systemic therapy at the time of screening, which is considered clinically significant by the Investigator.
14. Subject has a significant history of or ongoing chronic or recurrent infectious disease (e.g., infected indwelling prosthesis, osteomyelitis, chronic sinusitis), as determined by the Investigator.
15. Anticipating undergoing surgery or medical/dental procedure, receiving neuraxial anesthesia (spinal/epidural anesthesia), or undergoing spinal puncture during the study or within 7 days after study completion.
16. History of psychiatric disorders occurring within the last two years, which required the subject to be hospitalized or treated with medication.
17. Presence of a medical condition requiring regular treatment with prescription drugs (except hormonal contraceptives).
18. Use of pharmacologic agents or herbal products known to significantly induce or inhibit drug-metabolizing enzymes (especially inhibitors and inducers of CYP3A4 and P-gp such as ketoconazole, itraconazole, ritonavir, clarithromycin, rifampin, phenytoin, carbamazepine, St. John's Wort, etc.) within 30 days before initial dosing.
19. Use of drugs affecting hemostasis such as aspirin and other antiplatelet agents, other anticoagulants, heparin, thrombolytic agents, selective serotonin reuptake inhibitors (SSRIs), serotonin norepinephrine reuptake inhibitors (SNRIs), and nonsteroidal anti-inflammatory drugs (NSAIDs) within 14 days before initial dosing.
20. Receipt of any drug as part of a research study within 30 days before initial dosing.
21. Drug or alcohol addiction requiring treatment in the 12 months before initial dosing.
22. History of excessive alcohol consumption (on average more than 14 units of alcohol/week; 1 unit = 12 oz. beer, 6 oz. wine, 1 shot [1.5 oz.] of liquor) during the past 12 months.
23. Donation or significant loss of whole blood (480 mL or more) within 30 days or plasma within 14 days before initial dosing.
24. Positive test for HIV, Hepatitis B surface antigen or Hepatitis C antibody.
25. Positive test results for drugs of abuse or cotinine at screening.
26. If female, has a positive pregnancy test at screening.
27. Difficulty swallowing, as determined by the Investigator.
28. Use of tobacco- or nicotine-containing products within 1 year before initial dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Plasma Concentration (Cmax) of Apixaban under fasted condition | 0, 0.33, 0.67, 1.0, 1.5, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 8.0, 12.0, 16.0, 24.0, 36.0, 48.0 hours post dose
Area under the plasma concentration curve from time zero to last sampling time (AUC0-t) of Apixaban under fasted condition | 0, 0.33, 0.67, 1.0, 1.5, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 8.0, 12.0, 16.0, 24.0, 36.0, 48.0 hours post dose
Area under the plasma concentration curve from time zero to infinity (AUC0-∞) of Apixaban under fasted condition | 0, 0.33, 0.67, 1.0, 1.5, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 8.0, 12.0, 16.0, 24.0, 36.0, 48.0 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Philip Mathew, M.D., Principal Investigator — Novum Pharmaceutical Research Services, USA
Locations (1):
- Novum Pharmaceutical Research Services, Las Vegas, Nevada, United States